CLINICAL TRIAL: NCT02828709
Title: The Safety and Feasibility of Irreversible Electroporation for the Ablation of Small Renal Masses
Brief Title: Safety and Feasibility of IRE for SRMs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Prof. M.P. Laguna Pes (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Prof. M.P. Laguna Pes, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL5693501816
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irreversible electroporation (IRE) (Experimental): IRE is based on high current electric pulses, transferred between two or more placed needle electrodes. Charging the cell membrane causes holes in the cell membrane called "nanopores", resulting in increased permeability of the cell and subsequent cell death.
  Interventions: Device: Irreversible Electroporation

INTERVENTIONS:
Device: Irreversible Electroporation — Guided by CT and accompanied by an external spacer for fixation, needle electrodes will be placed. The amount of probes and probe placement will be attuned for specific tumour size and location, granting 15mm between the electrodes with an active tip length of 15mm. IRE pulses with pulse intensity of 1500 V/cm will be delivered in 90 consecutive pulses of 90µs.
  Other Names: Nanoknife

SUMMARY:
Irreversible Electroporation (IRE) is an emerging technique delivering electrical pulses to ablate tissue, with the theoretical advantage to overcome the main shortcomings of conventional thermal ablation. Recent short-term research showed that IRE for the ablation of renal masses is a safe and feasible treatment option. In an ablate and resect design, histopathological analysis 4 weeks after radical nephrectomy demonstrated that IRE targeted renal tumors were completely covered by ablation zone. In order to develop a validated long-term IRE follow-up study, it is essential to obtain clinical confirmation of the efficacy of this novel technology. Additionally, follow-up after IRE ablation obliges verification of a suitable imaging modality. The objectives of this study are the clinical efficacy and safety of IRE ablation of renal masses and to evaluate the use of cross-sectional imaging modalities in the follow-up after IRE in renal tumours.

This is a prospective, human, in-vivo study among 20 patients presenting with solid enhancing SRM on cross sectional imaging suspect for renal cell carcinoma (RCC). Preoperatively, imaging is required through Magnetic Resonance Imaging (MRI), Contrast-enhanced ultrasound (CEUS) and contrast-enhanced Computed Tomography (CT). Furthermore, serum creatinine levels and VAS scores are obtained. A biopsy of the SRM will be performed in preoperative setting. IRE ablation will be performed using CT-guidance and ablation success will be measured directly after the ablation through contrast-enhanced CT. Device related adverse events (AE) will be registered using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 guideline. One week post ablation only CEUS and MRI will be performed to limit exposure to ionizing radiation. At 3 months, 6 months and 12 months post ablation CEUS, MRI and CT will be performed. Additionally, at these time points serum creatinine levels and VAS scores will be obtained, and quality of life will be assessed through SF-36 questionnaires. Residual and recurrent disease will be assessed through tissue enhancement on cross sectional imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Solid, enhancing mass on cross sectional imaging
* Signed informed consent
* Candidate for focal ablative therapy

Exclusion Criteria:

* Irreversible bleeding disorders
* Inability/unwillingness to interrupt anticoagulation therapy
* Previous cryoablation, RFA or partial nephrectomy in affected kidney
* Anaesthesia Surgical Assignment (ASA), category ≤ IV
* ICD / pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
safety IRE ablation procedure (evaluating device and procedural adverse events using CTCAE v4.0) | 2 years
  To determine the safety and feasibility of IRE ablation of small renal masses (≤ 4cm), by evaluating device and procedural adverse events using CTCAE v4.0

SECONDARY OUTCOMES:
Clinical efficacy ((non-)presence of tumour enhancement on cross-sectional imaging post IRE) | 2 years
  To determine the clinical efficacy of IRE ablation of small renal masses (≤ 4cm), assessed by calculating recurrence and residual disease at follow-up, measured through the (non-)presence of tumour enhancement on cross-sectional imaging post IRE
Cross sectional imaging post ablation | 2 years
  To evaluate the use of CT, MRI, and CEUS in the imaging of ablation success, extend of the ablation zone, 1 week, 3 months, 6 months, and 1 year post IRE
Renal function | 2 years
  To evaluate the effect of RE ablation of small renal masses (≤ 4cm) on the renal function, measured by serum creatinine levels and estimated Glomerular Filtration Rate (eGFR)
Average length of hospital stay | 2 years
  To evaluate the effect of IRE ablation of small renal masses (≤ 4cm) on the length of hospital stay, measured in average stay in days
Quality of Life | 2 years
  To evaluate the effect of IRE ablation of small renal masses (≤ 4cm) on the quality of life, assessed through SF-36 questionnaires
Postoperative pain score | 1 year
  To asses the effect of IRE ablation of small renal masses (≤ 4cm), assessed through VAS score and analgesics use

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pilar Laguna Pes, MD, PhD, Principal Investigator — Academic Medical Center (AMC) Amsterdam
Locations (1):
- Academic Medical Center (AMC), Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomson KR, Cheung W, Ellis SJ, Federman D, Kavnoudias H, Loader-Oliver D, Roberts S, Evans P, Ball C, Haydon A. Investigation of the safety of irreversible electroporation in humans. J Vasc Interv Radiol. 2011 May;22(5):611-21. doi: 10.1016/j.jvir.2010.12.014. Epub 2011 Mar 25. PMID 21439847
- [Background] Wendler JJ, Ricke J, Pech M, Fischbach F, Jurgens J, Siedentopf S, Roessner A, Porsch M, Baumunk D, Schostak M, Kollermann J, Liehr UB. First Delayed Resection Findings After Irreversible Electroporation (IRE) of Human Localised Renal Cell Carcinoma (RCC) in the IRENE Pilot Phase 2a Trial. Cardiovasc Intervent Radiol. 2016 Feb;39(2):239-50. doi: 10.1007/s00270-015-1200-6. Epub 2015 Sep 4. PMID 26341653
- [Background] Trimmer CK, Khosla A, Morgan M, Stephenson SL, Ozayar A, Cadeddu JA. Minimally Invasive Percutaneous Treatment of Small Renal Tumors with Irreversible Electroporation: A Single-Center Experience. J Vasc Interv Radiol. 2015 Oct;26(10):1465-71. doi: 10.1016/j.jvir.2015.06.028. Epub 2015 Aug 4. PMID 26250855
- [Background] Pech M, Janitzky A, Wendler JJ, Strang C, Blaschke S, Dudeck O, Ricke J, Liehr UB. Irreversible electroporation of renal cell carcinoma: a first-in-man phase I clinical study. Cardiovasc Intervent Radiol. 2011 Feb;34(1):132-8. doi: 10.1007/s00270-010-9964-1. Epub 2010 Aug 15. PMID 20711837
- [Background] van den Bos W, de Bruin DM, van Randen A, Engelbrecht MR, Postema AW, Muller BG, Varkarakis IM, Skolarikos A, Savci-Heijink CD, Jurhill RR, Zondervan PJ, Laguna Pes MP, Wijkstra H, de Reijke TM, de la Rosette JJ. MRI and contrast-enhanced ultrasound imaging for evaluation of focal irreversible electroporation treatment: results from a phase I-II study in patients undergoing IRE followed by radical prostatectomy. Eur Radiol. 2016 Jul;26(7):2252-60. doi: 10.1007/s00330-015-4042-3. Epub 2015 Oct 8. PMID 26449559
- [Background] van den Bos W, Scheffer HJ, Vogel JA, Wagstaff PG, de Bruin DM, de Jong MC, van Gemert MJ, de la Rosette JJ, Meijerink MR, Klaessens JH, Verdaasdonk RM. Thermal Energy during Irreversible Electroporation and the Influence of Different Ablation Parameters. J Vasc Interv Radiol. 2016 Mar;27(3):433-43. doi: 10.1016/j.jvir.2015.10.020. Epub 2015 Dec 17. PMID 26703782
- [Background] Wagstaff PG, de Bruin DM, van den Bos W, Ingels A, van Gemert MJ, Zondervan PJ, Verdaasdonk RM, van Lienden KP, van Leeuwen TG, de la Rosette JJ, Laguna Pes MP. Irreversible electroporation of the porcine kidney: Temperature development and distribution. Urol Oncol. 2015 Apr;33(4):168.e1-7. doi: 10.1016/j.urolonc.2014.11.019. Epub 2014 Dec 31. PMID 25557146
- [Derived] Buijs M, van Lienden KP, Wagstaff PG, Scheltema MJ, de Bruin DM, Zondervan PJ, van Delden OM, van Leeuwen TG, de la Rosette JJ, Laguna MP. Irreversible Electroporation for the Ablation of Renal Cell Carcinoma: A Prospective, Human, In Vivo Study Protocol (IDEAL Phase 2b). JMIR Res Protoc. 2017 Feb 16;6(2):e21. doi: 10.2196/resprot.6725. PMID 28209559